CLINICAL TRIAL: NCT05435391
Title: A Prospective, Multicenter, Observational Diagnostic Study to Externally Validate an Artificial Intelligence 12-lead Electrocardiogram Analysis Algorithm to Detect Patients With Acute Myocardial Infarction Who Visit Emergency Medical Center
Brief Title: ROMIAE (Rule-Out Acute Myocardial Infarction Using Artificial Intelligence Electrocardiogram Analysis) Trial
Acronym: ROMIAE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: CHA University (Other)
Collaborators: Medical AI Co., Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: MAI-CRP-B0000
Record Dates: First submitted 2022-06-13; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-04

CONDITIONS: Myocardial Infarction or Chest Pain
Keywords: Deep Learning
MeSH Terms: conditions — Myocardial Infarction; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients with chest pain or who are clinically suspected as acute myocardial infarction with equivalent symptoms.

SUMMARY:
This study is a prospective multicenter observational study for external validation and model advancement of a deep learning based 12-lead electrocardiogram analysis algorithm targeting adult patients presenting to the emergency department with chest pain and acute myocardial infarction equivalent symptoms.

About 9,000 adult patients will be enrolled at 20 emergency medical centers in Korea. Artificial intelligence algorithms are manufactured by Medical AI Co., Ltd. It is an advanced version based on the model developed and published in 2020. It had the diagnostic performance of area under the receiver operating curve 0.901 and 0.951 for acute myocardial infarction and ST-segment elevation myocardial infarction, respectively. The primary endpoint is a diagnosis of acute myocardial infarction on the day of the emergency center visit, and the secondary endpoint is a 30-day major adverse cardiac event. From March 2022, patient registration will begin at centers that have been approved by the Institutional Review Board.

This is the first prospective multicenter emergency department validation study for a 12-lead electrocardiogram artificial intelligence algorithm to diagnose acute myocardial infarction. This study will give insight into the direction of future development by verifying whether the deep learning algorithm works well for patients visiting the real-world adult emergency medical center.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age with suspected chest pain and acute myocardial infarction
* The onset or worsening of the symptom occurs within 24 hours

Exclusion Criteria:

* Out-of-hospital cardiac arrest (OHCA): patients with sustained (>20 minutes) return-of-spontaneous-circulation are not excluded
* Patients in whom acute myocardial infarction can be clearly excluded, such as pneumothorax and traumatic chest pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 20 emergency departments in the Republic of Korea will participate in this study. These centers receive about 800,000 patients annually, and all of these hospitals are capable of their own emergency cardiovascular angiography and percutaneous coronary intervention.
Sampling Method: Non-Probability Sample
Enrollment: 8814 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of acute myocardial infarction (Type 1, 2) | Index admission
  Accuracy metrics include area under the receiver operating characteristics curve, sensitivity, specificity, positive predictive value, and negative predictive value, along with a 95% confidence interval.

SECONDARY OUTCOMES:
Major adverse cardiovascular event (MACE) | 30-day after index admission
  MACE is defined as death, myocardial infarction, stroke, target-vessel revascularization, or stent thrombosis occurring within 30 days of index visit. Accuracy metrics include area under the receiver operating characteristics curve, sensitivity, specificity, positive predictive value, and negative predictive value, along with a 95% confidence interval.

OTHER OUTCOMES:
AI ECG analysis versus clinical risk score (HEART score) | Index admission, 30-day after index admission
  HEART score is an acute coronary syndrome risk calculation tool introduced in recent guidelines, and consists of history, electrocardiogram, age, risk factor, and troponin. On a scale of 0 to 10, the higher the score, the higher the risk. Generally, a score of 7 or higher is classified as high risk. The prediction performance for the primary and secondary endpoints of the HEART score will be analyzed by comparing it with AI-ECG analysis.
AI ECG analysis versus clinical risk score (GRACE 2.0 score) | Index admission, 30-day after index admission
  GRACE 2.0 score is a tool for estimating short- and long-term risk in acute coronary syndrome. A low score indicates low risk, and a high score indicates a high risk group. Based on recent guidelines, patients with acute coronary syndrome are categorized as low (≤108 GRACE score), medium (109-140 GRACE score) and high risk (>140 GRACE score). The prediction performance for the primary and secondary endpoints of the GRACE 2.0 score will be analyzed by comparing it with AI-ECG analysis.
AI ECG analysis versus cardiac biomarker | Index admission
  The performance of cardiac biomarker (hs-troponin I or T) for the diagnosis of acute myocardial infarction during index visit will be compared with AI ECG analysis diagnostic performance.
AI ECG analysis versus physician's ECG score | Index admission
  The attending physician determines a score between 0 and 10 for the probability of acute myocardial infarction based on the results of the initial patient assessment and the first 12-lead ECG. A score of 0 indicates that the probability of acute myocardial infarction is 0%, and a score of 10 indicates a probability of 100%. The diagnostic performance of this score for acute myocardial infarction will be compared with AI ECG analysis.

CONTACTS AND LOCATIONS:
Overall Officials: KS Kim, MD, PhD, Principal Investigator — CHA University School of Medicine
Locations (1):
- CHA Bundang Medical Center, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shin TG, Lee Y, Kim K, Lee MS, Kwon JM; ROMIAE study group. ROMIAE (Rule-Out Acute Myocardial Infarction Using Artificial Intelligence Electrocardiogram Analysis) trial study protocol: a prospective multicenter observational study for validation of a deep learning-based 12-lead electrocardiogram analysis model for detecting acute myocardial infarction in patients visiting the emergency department. Clin Exp Emerg Med. 2023 Dec;10(4):438-445. doi: 10.15441/ceem.22.360. Epub 2023 Nov 28. PMID 38012820